CLINICAL TRIAL: NCT01053559
Title: Open Label Investigator Initiated, Single Site Study of Mucosal Healing in Patients With Small Bowel Crohn's Disease Treated With Certolizumab Pegol (Cimzia) Assessed by Wireless Capsule Endoscopy
Brief Title: Assessment of Small Bowel Healing in Crohn's Disease Patients Treated With Cimzia Using Wireless Capsule Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shafran Gastroenterology Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Ira Shafran M.D., Principal Investigator, Shafran Gastroenterology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exempt IND
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- certolizumab pegol (Other): Subjects will receive FDA approved Cimzia injections as indicated on the product label. Subjects will undergo 3 wireless capsule endoscopies, one at screening,Day 84 and Day 168 as well as monthly bloodwork.
  Interventions: Drug: certolizumab pegol

INTERVENTIONS:
Drug: certolizumab pegol — 400mg subcutaneous injections at week 0, week 2, week 4, then every 4 weeks thereafter
  Other Names: Cimzia

SUMMARY:
Wireless Capsule Endoscopy has been the most reliable diagnostic standard for small bowel Crohn's disease. Endoscopic healing is an important endpoint to measure response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 with confirmed Crohn's disease that includes small bowel disease
* Moderately to severely active disease (CDAI score >220 and < 450)
* Stable doses of steroids, 5-ASA, antibiotics, Immunosuppressants

Exclusion Criteria:

* Any and all contraindications to the use of certolizumab pegol (including but not limited to hepatitis, infection, abscess, malignancy, congestive heart failure [CHF], cytopenia)
* Small bowel obstruction, stricture, or any contraindication for capsule endoscopy
* Previous treatment with certolizumab pegol
* Are pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mucosal Healing | 180 Days

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) Level | 180 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shafran, M.D., Principal Investigator — Shafran Gastroenterology Center
Locations (1):
- Shafran Gastroenterology Center, Winter Park, Florida, United States

REFERENCES:
- See also: Practice Website — http://www.shafran.net